CLINICAL TRIAL: NCT02394990
Title: A Randomised Controlled Trial to Evaluate a Violence Brief Intervention (VBI) for Adult Male Patients With Facial Injuries Sustained as a Result of Interpersonal Violence
Brief Title: Violence Brief Intervention Pilot v1.1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GN14NU421
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Alcohol Consumption; Violence; Facial Injuries
MeSH Terms: conditions — Alcohol Drinking; Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Violence Brief Intervention (Experimental): Participants receive a standard of care brief motivational intervention (BMI) to address alcohol consumption (ABI) based on self reported use and their relationship between consumption and behavior, followed by an additional BMI to address how involvement in violence (VBI) impacts their life, relationship to social norms, and strategies to avoid violence.
  Interventions: Behavioral: Violence Brief Intervention
- Control (Active Comparator): Participants receive only ABI
  Interventions: Behavioral: ABI

INTERVENTIONS:
Behavioral: Violence Brief Intervention — Strategies for self assessment of consequences of violent behavior and strategies for avoidance of violence
  Other Names: VBI
  Arms: Violence Brief Intervention
Behavioral: ABI
  Arms: Control

SUMMARY:
This study is a randomised controlled trial of a new brief intervention with young (16-29) adult male patients who have a facial injury sustained as a result of interpersonal violence (fighting or assaults). It will be undertaken at the Maxillofacial outpatient trauma clinic at the Southern General Hospital, Glasgow. The major risk factors associated with facial injury in Scotland are male gender, young age, interpersonal violence and alcohol. Previous research with facial injury patients attending this clinic has shown that an Alcohol Brief Intervention (ABI) is effective in helping reduce alcohol consumption, so all patients are now offered ABI as standard practice. ABI is delivered by trained nurses from Addiction Services. This will not be withdrawn. In addition we wish to offer some patients a Violence Brief Intervention (VBI). This will be delivered by the same nurses who deliver the ABI. The study is randomised so only those selected at random will receive this extra intervention and all others will receive treatment as normal (ABI only). VBI is a short psychological intervention which uses Brief Motivational Interviewing (BMI) to encourage reflection of involvement in violence and consideration of strategies to avoid future violence. The intervention also compares participants' attitudes towards violence to those of their peers. The intervention takes about 15 minutes, and patients will be involved for an additional 30-45 minutes longer than normal when they attend the clinic, including consent and baseline data collection. Patients will be followed up by telephone at 1, 3 and 6 months, and asked a suite of questions which will take approximately 15 minutes on each occasion. We wish to determine whether a VBI of this type has any effect on attitudes to violence or propensity for involvement in violence or on reinjury, examined through self report measures and routinely collected health and criminal justice data at 12 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* facial trauma patients
* Facial injury resulting from interpersonal violence (whether victim or perpetrator)
* Able to give informed consent
* Willing to commit to screening intervention and follow up programme lasting 6 months
* Within 28 days of injury
* Willing to provide either a contact telephone number or email address for the followup surveys
* Participants score ≥ 3/16 on the Fast Alcohol Screening Test (FAST)

Exclusion Criteria:

* Unable to give informed e.g. adults with dementia, severe psychiatric problems, patients with learning difficulties who cannot consent for themselves
* Under 16 or over 29 years of age.
* Injury more than 28 days old
* Participants score ≤ 2/16 on the FAST measure

Ages: 16 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Re-admission for trauma injury | 12 months post-intervention
Named in police crime report as perpetrator, victim or witness of violence | 12 months post-intervention
Attitudes toward violence | 1, 3 and 6 months post intervention

SECONDARY OUTCOMES:
Participant relationships to alcohol measured using the Fast Alcohol screening test | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christine Goodall, BDS, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Department of Oral and Maxillofacial Surgery, Southern General Hospital, Glasgow, United Kingdom